CLINICAL TRIAL: NCT05057936
Title: Antibody Response After COVID-19 Vaccination in Chronic Kidney Disease and Kidney Transplant Patients
Brief Title: Antibody After COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Other Study IDs: 101/64
Record Dates: First submitted 2021-09-23; First posted 2021-09-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Breakthrough Infection; CKD; Kidney Transplant; Vaccination
Keywords: COVID-19; vaccine; Neutralising antibody; chronic kidney disease; kidney transplant; anti-spike RBD IgG; nucleocapsid antibody; interferon gamma
MeSH Terms: conditions — COVID-19; Breakthrough Infections; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: Healthy healthcare workers
  Interventions: Biological: COVID vaccine
- Chronic kidney disease (CKD): CKD stage 3-5 (eGFR < 60 mL/min/1.73m3)
  Interventions: Biological: COVID vaccine
- Dialysis patients: CKD stage 5 requiring HD
  Interventions: Biological: COVID vaccine
- kidney transplant patients: patients receiving kidney transplantation for more than 3 months
  Interventions: Biological: COVID vaccine
- dialysis patients: CKD patients requring continuos ambulatory peritoneal dialysis
  Interventions: Biological: COVID vaccine

INTERVENTIONS:
Biological: COVID vaccine — The enrolled patients will received COVID-19 vaccine according to the vaccine protocol in Thailand ie The ChAdox-1 nCOV-19 vaccine (day 1, day 84, 12 weeks duration) or Corona vac 2 doses (day 2, day 21, 3 weeks duration) of the study. All the participants underwent blood drawn for antibody and cellular immunity measurement before the final dose of vaccination, with 7 days before first vaccine dose and eight weeks after the second doses

SUMMARY:
Chronic kidney disease (CKD) including patients on dialysis and kidney transplant recipients. represents the special subgroups of patients that required protection during the Severe Coronavirus Disease 2019 (COVID-19) pandemic .Since COVID-19 is associated with severe morbidity and mortality in these particular subgroup of patients, the main strategies is proper and rapid vaccination. CKD patients usually have a reduced immune responses, vaccination in these group of patients usually require higher dosage and more frequent dose since the vaccine response is short-lived and less response especially in dialysis patients5 .In patients with normal renal function,the immunity is durable but with modest declines at 6-8months. One study showed a linear decline in IgG in dialysis patients for up to 3months , but there are otherwise limited data.

Previous reports of the vaccination in CKD patient involved mainly the mRNA vaccines. The recent reports of seroconversion rate dialysis patients receiving two doses of BNT 162b2 vaccine (Pfizer BioNtech) was lower than in control. In Thailand, the main vaccines available are Coronavac (Sinovac Life Science, Beijing, China) and ChadOx1 nCoV-19 (Oxford-Astra Zeneca) which was dispensed all over the country since April 2021. Data of the efficacy and safety of these vaccines in these patient groups is lacking. Therefore, the aim of this study is to measure the antibody and cellular responses in CKD patients including those with dialysis therapy and kidney transplantation and monitor the adverse events after the first and second doses of after vaccination. The incidence rate of Sars-COV2 infection post vaccination was also observed.

DETAILED DESCRIPTION:
This is a prospective cohort study that included 4 different cohorts i.e CKD ,hemodialysis ( HD), continuous ambulatory peritoneal dialysis (CAPD) , kidney transplant (KT) patients and a control group without kidney failure at Faculty of Medicine, Vajira Hospital,Navamindradhiraj University from June -December 2021. The inclusion criteria were CKD stage 3-5 (eGFR < 60 mL/min/1.73m3), CKD patients receiving HD,CAPD and KT. The participants of the healthy control group consists of volunteer health care workers who had been vaccinated according to the nation vaccination schedule. Participants in both groups needed to be 18-90 years old. The exclusion criteria were allergy to the components of vaccines, unable to receive the vaccine according to the schedule,fever or concomitant serious illnesses and had side effect from the first dose of vaccination. Patients or individuals with prior COVID-19 infection in the past (diagnosed via patients history and serological test for nucleocapsid (NCP) antibody were excluded from the study. The study protocol was approved by the local Ethics Committed and participants were enrolled after written informed consent was obtained. The study who performed in accordance with the principles of the Declaration of Helsinki and Good Clinical Practice. The vaccine used was authorized by the Thai Food and Drug Administration and the Department of Medical Sciences (DMS).

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3-5 (eGFR < 60 mL/min/1.73m3)
* CKD stage 5 patients receiving HD,CAPD and KT for more than 3 months.
* The participants of the healthy control group consists of volunteer health care workers who had been vaccinated according to the nation vaccination schedule

Exclusion Criteria:

* allergy to the components of vaccines
* unable to receive the vaccine according to the schedule
* fever or concomitant serious illnesses
* had side effect from the first dose of vaccination
* prior COVID-19 infection in the past (diagnosed via patients history and serological test for nucleocapsid (NCP) antibody

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD stage 3-5 and those require renal replacment therapy with HD,CAPD or Kidney trasnplantation
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity after COVID-19 vaccination | Baseline before vaccination
  levels of SARS-CoV2 spike S1-specific immunoglobulin (IgG) antibody concentration
Immunogenicity after COVID-19 vaccination | The second dose of vaccination
  levels of SARS-CoV2 spike S1-specific immunoglobulin (IgG) antibody concentration
Immunogenicity after COVID-19 vaccination | Eight weeks after the second dose of vaccination
  levels of SARS-CoV2 spike S1-specific immunoglobulin (IgG) antibody concentration
Immunogenicity after COVID-19 vaccination | Baseline before vaccination
  Viral neutralization test measured by surrogate virus neutralization test (SVNT)
Immunogenicity after COVID-19 vaccination | The second dose of vaccination
  Viral neutralization test measured by surrogate virus neutralization test (SVNT)
Immunogenicity after COVID-19 vaccination | Eight weeks after the second dose of vaccination
  Viral neutralization test measured by surrogate virus neutralization test (SVNT)
Immunogenicity after COVID-19 vaccination | Baseline before vaccination
  Cellular immunity by interferon gamma level
Immunogenicity after COVID-19 vaccination | The second dose of vaccination
  Cellular immunity by interferon gamma level
Immunogenicity after COVID-19 vaccination | Eight weeks after the second dose of vaccination
  Cellular immunity by interferon gamma level

SECONDARY OUTCOMES:
rates of adverse events after vaccination | 28 days
  drug allergy ,skin rash,liver toxicity
the incidence of COVID-19 breakthrough infection after vaccination | 28 days
  number of cases that develop COVID-19 infection after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine,Vajira Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The data that present in this study will be deposited in Mendeley osother data repository sited as appropriate
Supporting Information: Study Protocol, SAP
Time Frame: after publication is accepted and indefinitely
Access Criteria: additional data related to this paper may be requested from the corresponding author

REFERENCES:
- [Background] Hilbrands LB, Duivenvoorden R, Vart P, Franssen CFM, Hemmelder MH, Jager KJ, Kieneker LM, Noordzij M, Pena MJ, Vries H, Arroyo D, Covic A, Crespo M, Goffin E, Islam M, Massy ZA, Montero N, Oliveira JP, Roca Munoz A, Sanchez JE, Sridharan S, Winzeler R, Gansevoort RT; ERACODA Collaborators. COVID-19-related mortality in kidney transplant and dialysis patients: results of the ERACODA collaboration. Nephrol Dial Transplant. 2020 Nov 1;35(11):1973-1983. doi: 10.1093/ndt/gfaa261. PMID 33151337
- [Background] Kengibe PY, Makulo JR, Nlandu YM, Lepira FB, Sumaili EK, Bukabau JB, Mbendi CN, Ahuka SM, Tshimpi AW, Ngoma PK, Mangani NN, Mbendi SN. Response to single dose hepatitis B vaccine in Congolese non-HIV hemodialysis patients: a prospective observational study. Pan Afr Med J. 2019 Oct 31;34:122. doi: 10.11604/pamj.2019.34.122.19603. eCollection 2019. PMID 33708291
- [Background] Bensouna I, Caudwell V, Kubab S, Acquaviva S, Pardon A, Vittoz N, Bozman DF, Hanafi L, Faucon AL, Housset P. SARS-CoV-2 Antibody Response After a Third Dose of the BNT162b2 Vaccine in Patients Receiving Maintenance Hemodialysis or Peritoneal Dialysis. Am J Kidney Dis. 2022 Feb;79(2):185-192.e1. doi: 10.1053/j.ajkd.2021.08.005. Epub 2021 Sep 8. PMID 34508833
- [Background] Carr EJ, Kronbichler A, Graham-Brown M, Abra G, Argyropoulos C, Harper L, Lerma EV, Suri RS, Topf J, Willicombe M, Hiremath S. Review of Early Immune Response to SARS-CoV-2 Vaccination Among Patients With CKD. Kidney Int Rep. 2021 Sep;6(9):2292-2304. doi: 10.1016/j.ekir.2021.06.027. Epub 2021 Jul 6. PMID 34250319
- [Background] Grupper A, Sharon N, Finn T, Cohen R, Israel M, Agbaria A, Rechavi Y, Schwartz IF, Schwartz D, Lellouch Y, Shashar M. Humoral Response to the Pfizer BNT162b2 Vaccine in Patients Undergoing Maintenance Hemodialysis. Clin J Am Soc Nephrol. 2021 Jul;16(7):1037-1042. doi: 10.2215/CJN.03500321. Epub 2021 Apr 6. PMID 33824157
- [Background] Labriola L, Scohy A, Seghers F, Perlot Q, De Greef J, Desmet C, Romain C, Morelle J, Yombi JC, Kabamba B, Rodriguez-Villalobos H, Jadoul M. A Longitudinal, 3-Month Serologic Assessment of SARS-CoV-2 Infections in a Belgian Hemodialysis Facility. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):613-614. doi: 10.2215/CJN.12490720. Epub 2020 Nov 18. No abstract available. PMID 33208402
- [Background] Ikizler TA, Coates PT, Rovin BH, Ronco P. Immune response to SARS-CoV-2 infection and vaccination in patients receiving kidney replacement therapy. Kidney Int. 2021 Jun;99(6):1275-1279. doi: 10.1016/j.kint.2021.04.007. Epub 2021 Apr 20. PMID 33931226
- [Background] Torreggiani M, Blanchi S, Fois A, Fessi H, Piccoli GB. Neutralizing SARS-CoV-2 antibody response in dialysis patients after the first dose of the BNT162b2 mRNA COVID-19 vaccine: the war is far from being won. Kidney Int. 2021 Jun;99(6):1494-1496. doi: 10.1016/j.kint.2021.04.010. Epub 2021 Apr 20. No abstract available. PMID 33887320
- [Background] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298